CLINICAL TRIAL: NCT04353648
Title: Assessment of Muscle Metabolic Phenotype by the Use of Point-of-care MSK Ultrasound Imaging.
Brief Title: Assessing Muscle Metabolic Phenotype by MSK Ultrasound
Status: Terminated | Type: Observational
Why Stopped: Insufficient staff
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103143
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Ultrasound; CT; MuscleSound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Duke ICU/Trauma Center Patients: Any patient admitted to the Duke Trauma Center or Duke ICU will be approached to participate in this study.

SUMMARY:
The purpose of this study is to test whether ultrasound images (pictures) can be used as a valid assessment of muscle quality in different muscle groups during Intensive Care stay. This new approach would allow clinicians to obtain frequent skeletal muscle images and would enable doctors to observe any changes over time in muscle quality that could occur during ICU stay.

Participants in this study will have ultrasound images made of their leg-, chest- and jaw muscles taken on every day until ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* admission Duke Trauma center, SICU, MICU, or CT ICU
* >18 years of age

Exclusion Criteria:

* <18 years of age
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to a Duke Trauma center, SICU, MICO, or CT ICU
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Muscle Quality from the rectus femoris, vastus lateralis, intermedius, intercostalis, temporalis and styloglossus | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  Ultrasound-derived area of intramuscular adipose tissue (IMAT) and intramuscular glycogen content from the rectus femoris, vastus lateralis, intermedius, intercostalis, temporalis and styloglossus
Muscle volume and thickness from the rectus femoris, vastus lateralis, intermedius, intercostalis, temporalis and styloglossus | Minimum of every other day while in ICU (up to 10 days). Once discharged from ICU minimum of 3x a week until discharge (up to 3 weeks)
  Ultrasound-derived volume and thicknessfrom the rectus femoris, vastus lateralis, intermedius, intercostalis, temporalis and styloglossus

SECONDARY OUTCOMES:
Changes of Intramuscular adipose tissue (IMAT) content and muscle volume/thickness from the psoas at the Level of L3/L4 | Up to 1 year
  the change over time of (standard of care) CT-derived area of intramuscular adipose tissue in cm2
Changes of Intramuscular adipose tissue (IMAT) content and muscle volume/thickness from the intercostal muscle at the Level of Th3/Th4 | Up to 1 year
  the change over time of (standard of care) CT-derived area of intramuscular adipose tissue in cm2
Changes of Intramuscular adipose tissue (IMAT) content and muscle volume/thickness from the intercostal muscle at the Level of the head | Up to 1 year
  the change over time of (standard of care) CT-derived area of intramuscular adipose tissue in cm2

CONTACTS AND LOCATIONS:
Overall Officials: Paul Wischmeyer, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No